CLINICAL TRIAL: NCT02258568
Title: Postnatal Smoking Relapse, Its Associated Risk Factors, and a Proactive Sustainable Preventive Intervention
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Cristian Ioan Meghea, Scientific Researcher, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PN-II-RU-TE-2012-3-0209
Record Dates: First submitted 2014-09-29; First posted 2014-10-07 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Cigarette Smoking
Keywords: Cigarette Smoking; Pregnancy; Postpartum smoking relapse; Romania
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking abstinence counseling (Experimental): Telephone motivational counseling sessions supporting smoking abstinence
  Interventions: Behavioral: Smoking abstinence counseling
- Control (No Intervention): Do not receive telephone motivational counseling sessions supporting smoking abstinence

INTERVENTIONS:
Behavioral: Smoking abstinence counseling — Telephone smoking abstinence counseling based on motivational interviewing concepts
  Arms: Smoking abstinence counseling

SUMMARY:
This study will assess the extent of postpartum smoking relapse among Romanian women, the associated risk factors, and will develop, implement, and pilot-test a randomized trial smoking relapse intervention incorporating innovative research concepts in a social and cultural acceptable manner. The primary hypothesis is that the intervention will increase mothers' smoking abstinence rates.

DETAILED DESCRIPTION:
Overview.

This four-year longitudinal project will enroll a total of 425 women who spontaneously quit smoking during pregnancy. The recruitment will take place during the delivery hospital stay in two of the largest obstetric-gynecology hospitals in Cluj-Napoca, Romania. The investigators will design, pre-test (Objective 1), apply, and evaluate a postpartum smoking relapse preventive randomized intervention among the first 250 recruited women and their husbands (Objective 2): 125 couples in the intervention group and 125 couples in the control group, comparing the women's relapse rates at 6 months postpartum. The project will continue to enroll and follow-up 175 additional women for a total of 300 not subjected to the intervention (125+175) to assess the extent of postpartum smoking relapse and associated risk factors in a prospective cohort study (Objective 3).

The work plan.

The first 6 months of the project consisted of a preparatory phase. Objective 1 was completed in the first 9 months of the project, and milestones included focus groups, interviews with women, their husbands, and medical staff, the design of the intervention and pre-testing its acceptability. Objective 2 is completed between months 10-24 of the project. Milestones include: recruiting 250 couples (months 10-30), applying the intervention (months 10-33), the follow-up assessment (months 16-36), and preliminary analyses (months 13-36). Objective 3 is completed between months 19-45 of the project. Milestones include: recruiting 175 additional women (months 19-39), the follow-up assessment (months 25-45), and preliminary analyses (months 22-45). The last 12 months (months 37-48) of the project will be used to conclude the project, including finalizing the database and analyses, preparing a final report, and preparing articles for publication.

Objective 1: Design, pre-test, and refine an innovative intervention for preventing smoking relapse after pregnancy to maximize feasibility and potential impact.

This objective represented the qualitative developmental phase of the postpartum relapse intervention in order to tailor the intervention to the needs of the target population. The focus-groups and interviews aimed to qualitatively explore the issues related to the women's motivation and self-efficacy, the two key components of the planned intervention. To develop the postpartum smoking relapse intervention strategy the Motivation and Problem Solving (MAPS) strategy of Reitzel and colleagues was followed, the newest approach in the relapse prevention field, incorporating both motivational and self-efficacy components into the intervention, adapted to local attitudes and preferences. MAPS was successful in preventing relapse. The intervention is based on Motivational Interviewing and the seminal relapse prevention model, probably the most prominent theory of smoking cessation and relapse. Self-efficacy is viewed as the principal causal determinant of successful abstinence, among other individual and contextual factors, is hypothesized to increase. The model also specifies that the individual needs to be sufficiently motivated to avoid relapse. Briefly, the phone counseling sessions consist of information about the benefits of abstinence to increase motivation, and helping women identify and manage high-risk relapse situations, therefore enhancing their self-efficacy. The aim is to deliver consistent repeated advice by a trained professional over the phone in the postpartum period. Following the newest approaches in the field, the smoking husbands/partners are also targeted with brief motivational advice using the birth as a teachable moment to quit. Two psychologists were trained to deliver the phone motivational advice. Self help materials were also created and are distributed to all 250 women participating in the trial. A randomization algorithm was set up to assign patients into the intervention or control groups.

Objective 2: Implement and evaluate an intervention to prevent maternal smoking relapse after pregnancy in a randomized controlled trial setting.

Participants. The aim is to recruit 250 pre-randomized (125 intervention vs. 125 control group) mothers at birth who quit smoking in the 2 months before pregnancy or no later than the end of 1st pregnancy trimester and remained abstinent until delivery, biochemically confirmed through expired carbon monoxide. The mothers are approached during the delivery hospital stay in two of the largest obstetrics-gynecology clinics in Cluj-Napoca, Romania. Enrollment criteria include willingness and ability to participate in the study, age 18 or older, married or living with a stable partner, with a mobile phone, and willing to provide mobile phone contact for their husband or partner. Their husband or life partner is also approached and invited into the study at recruitment, if present, or by phone in the first weeks after birth.

Procedures. At enrollment, all 250 participants are given self-help materials and 5-10 min of brief advice offered by the trained research personnel consisting of encouragement to remain quit, and a review of the smoking risks and the benefits of abstinence. The mothers in the intervention group additionally receive three telephone-based counseling sessions delivered by trained professionals over the phone at 1 week, 1 month, and 3 months after birth. All smoking husbands or partners of the mothers in the intervention group are contacted in the first weeks after birth and are offered one phone motivational session to quit and support their wife's abstinence. To incentivize the couples to remain in the study and to appreciate their time and effort, gift certificates are mailed for baby-related merchandise around the 1-month and 6-month follow-up contacts.

Outcomes. The project follows-up with the couples at 6 months postpartum. Postpartum maternal abstinence is the main outcome, defined as maintaining smoke-free status continuously until the 6-month follow-up. The postpartum maternal abstinence is biochemically verified through expired carbon monoxide (CO) at 6-months postpartum (CO) <10 ppm. Secondary outcomes of interest are the maternal number of cigarettes smoked, self-efficacy, and motivation. The self-reported smoke status of the husband/partner is another outcome of interest.

Maternal characteristics. An extended prenatal questionnaire is used at recruitment and at the 6-month follow-up. Based on the prior literature on the predictors of postpartum relapse, the questionnaire includes demographics (such as age, education, and ethnicity), health history (prior pregnancies history, contraception use and feelings about the pregnancy), mental health (depressive symptoms, stress, anxiety), nicotine dependence before quitting, an extensive section on smoking knowledge and attitudes, other substance use, breast feeding, and having a life partner who smokes (as reported by the new mother).

Analytical plan. The required sample (100 intervention vs. 100 control at final follow-up) was calculated assuming abstinence rates of 0.3-0.4 (70% or 60% relapse) in the control group compared to anticipated 0.5-0.6 in intervention group, in order to attain 80% statistical power to detect the difference in two-tailed comparisons, alpha 0.05. Beginning with 125 couples in the intervention vs. 125 in the control group at enrollment, consistent with prior projects in Romania, 20% attrition is assumed by the final follow-up at 6 months after birth (100 vs. 100). To evaluate the effectiveness of the intervention, initially unadjusted comparisons of the outcomes in intervention vs. the control groups will be performed. Regression analyses will be used to adjust for group dissimilarities when differences have p-values less than 0.10. A cost-benefit analysis of the intervention will also be performed. The intervention costs will be compared to the health benefits derived from increased mother abstinence rates, increased father quit rates, and reduced family exposure to tobacco smoke. The health benefits will be monetized using estimates available in the research literature. In addition, economic analyses will be presented for various scenarios in which the proposed intervention can be integrated and sustained in the existing Romanian health system.

Objective 3. Assess the extent of postpartum smoking relapse and associated risk factors among women who spontaneously quit smoking during pregnancy.

Participants. To assemble a larger sample of women who quit smoking during pregnancy, 175 additional women are recruited during the delivery hospital stay, for a total of 300 (125 from Objective 2 + 175) women not subjected to the intervention. For consistency, they are offered the same self-help materials, brief advice, and gift certificate incentives (see Objective 2).

Outcomes and maternal characteristics. Postpartum maternal abstinence at 6 months postpartum are the main outcome of interest. A secondary outcome of interest is the maternal number of cigarettes smoked postpartum. Associations with all the maternal characteristics described above will be explored(see Objective 2), with a particular focus on the mental health, the nicotine dependence before quitting, breast feeding, and having a partner who smokes.

Analytical plan. Descriptive and multivariate analyses will be used to compare the women who relapse to the ones who remain abstinent. Descriptive analyses (counts and percentages) will assess the extent of postpartum smoking relapse and explore unadjusted associations between various characteristics and risk factors of the women and their postpartum smoking status: abstinent vs. relapsed. Multivariate logistic analyses will uncover the independent, adjusted, effects of individual and interacted factors, statistically adjusting for the effects of all other variables included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to participate in the study
* Married or living with a stable partner
* Mobile phone
* Willing to provide mobile phone contact for their husband or partner

Exclusion Criteria:

* Age<18 (minor age in Romania)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Postpartum maternal smoking abstinence | 6 months postpartum
  Defined as maintaining smoke-free status continuously until the 6-month follow-up. The postpartum maternal abstinence will be biochemically verified through expired carbon monoxide (CO) at 6-months postpartum

SECONDARY OUTCOMES:
Maternal number of cigarettes smoked | 6 months postpartum
Maternal self-efficacy scores on the Romanian version of the General Self Efficacy scale | 6 months postpartum
Maternal motivation scores on the Reasons for Quitting scale | 6 months postpartum
Self-reported smoke status of the husband/partner. | 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Cristian I Meghea, PhD, Principal Investigator — Michigan State University
Locations (1):
- Cluj School of Public Health, Cluj-Napoca, Cluj, Romania